CLINICAL TRIAL: NCT04589923
Title: The Measurement of VItal SIgns by Lifelight® Data Collect Software in comparisON to the Standard of Care in Acutely Unwell Patients - The VISION-Acute Study
Brief Title: The VISION-Acute Study
Status: Completed | Type: Observational
Sponsor: Xim Limited (Industry)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government); Mind Over Matter Medtech Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PHT/2020/50
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hypertension; Hypoxia; Hypotension
Keywords: vital signs; innovation; lifelight; blood pressure; oxygen saturation; contactless; COVID-19; rPPG
MeSH Terms: conditions — Hypertension; Hypoxia; Hypotension; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - participants expected to have abnormal oxygen saturation: Within each study session, participants will have their oxygen saturation, heart rate and respiratory rate measured three times using standard of care equipment and methods. At the same time, video of the participant's face will be captured using the Lifelight® Data Collect app running on a tablet positioned opposite them. The app will upload the RGB data extracted from this video to the cloud for subsequent analysis and processing aligned to the study's primary and secondary objectives only. The app does not return any measurements to the user or participant.
  Interventions: Device: Lifelight® Data Collect Oxygen Saturation Group
- Group 2 - participants expected to have abnormal blood pressure: Within each study session, participants will have their blood pressure and respiratory rate measured three times using standard of care equipment. At the same time, video of the participant's face will be captured using the Lifelight® Data Collect app running on a tablet positioned opposite them. The app will upload the RGB data extracted from this video to the cloud for subsequent analysis and processing aligned to the study's secondary objectives only. The app does not return any measurements to the user or participant.
  Interventions: Device: Lifelight® Data Collect Blood Pressure Group

INTERVENTIONS:
Device: Lifelight® Data Collect Blood Pressure Group — The staff member will prepare for and take the participant's routine observations using standard clinical equipment during the same 60-second period that video is captured of the participant's face using Lifelight® Data Collect (from which only the RGB data will be uploaded to the cloud). These measurements and RGB data capture will be repeated two times following the initial observations. Once measurements are concluded, the study staff member will complete the post-measurement observation questions.
  Groups: Group 2 - participants expected to have abnormal blood pressure
Device: Lifelight® Data Collect Oxygen Saturation Group — The staff member will prepare for and take the participant's routine observations using standard clinical equipment during the same 60-second period that video is captured of the participant's face using Lifelight® Data Collect (from which only the RGB data will be uploaded to the cloud). These measurements and RGB data capture will be repeated two times following the initial observations. Once measurements are concluded, the study staff member will complete the post-measurement observation questions.
  Groups: Group 1 - participants expected to have abnormal oxygen saturation

SUMMARY:
AIM: We propose an innovative approach using Lifelight® smart technology that will enable the continued provision of high level patient care at the same time as reducing pressure on nursing and equipment resources.

METHOD : Lifelight® is a computer program ("app") which can be used on smart devices that contain a camera. It is able to measure all of the vital signs by measuring very small changes in skin colour that occur each time the heart beats. This means that it does not need to touch the patient. We believe this could be an effective way of measuring vital signs, especially during the COVID-19 pandemic when prevention of cross-contamination between patients is essential. Patients are also likely to be reassured by a contactless approach.

During this study, we will recruit two groups of people who are hospitalised with an acute illness. The first group will be people expected to have abnormal blood oxygen levels such as those with acute respiratory problems including those with COVID-19. The second group will be people expected to have abnormal blood pressure. These Lifelight vital signs will be compared to measurements from standard clinical equipment.

The exact number of participants recruited will depend on how quickly the app "learns" and how many of the vital signs collected are outside of the normal range. For the first group of participants, we will use a camera to collect data about the changes in their face and use this to teach the app how to measure blood oxygen level and also to check how well the app measures blood oxygen level, heart rate and respiratory rate. For the second group of participants, we will use a camera to collect data about the changes in their face to check how well the app measures blood pressure and respiratory rate. All of the data will be kept secure and participants will not be able to be identified.

DETAILED DESCRIPTION:
Following informed consent, the study staff member will complete a very brief set of demographic and medical history questions, limited to the presence or absence of medical problems and treatment for them.

Participants will be recruited into either Group 1 or Group 2 depending on their previous clinical observations assessed during screening.

* Group 1 participants will have oxygen saturation, heart rate and respiratory rate measured.
* Group 2 participants will have blood pressure and respiratory rate measured.

For all participants, the study team will complete a set of pre-measurement observation questions. Background luminosity will be measured using a handheld lux meter. The staff member will then prepare for and take the participant's routine observations using standard clinical equipment during the same 60-second period that video is captured of the participant's face using Lifelight® Data Collect (from which only the RGB data will be uploaded to the cloud). These measurements and RGB data capture will be repeated two times following the initial observations. Once measurements are concluded, the study staff member will complete the post-measurement observation questions.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years old
2. Requiring hospital admission with an acute illness
3. Potential for vital signs to be outside of the normal ranges on the basis of their clinical status

Exclusion Criteria:

1. Participants unable to undertake simultaneous blood pressure monitoring in both arms will be excluded from Group 2, for example participants with an arterio-venous fistula for dialysis or in cases of lymphoedema following breast cancer surgery
2. Participants admitted to Intensive Care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients - adults
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2022-05-07 (Actual)

PRIMARY OUTCOMES:
Primary Objective | 3 months
  Train Lifelight® oxygen saturation algorithms with hypoxic individuals.

SECONDARY OUTCOMES:
Secondary Objective 1 | 3 months
  Measure oxygen saturation using Lifelight® with accuracy closer to +/- 4%.
Secondary Objective 2 | 3 months
  Measure heart rate using Lifelight® with accuracy closer to RMSE of 3bpm.
Secondary Objective 3 | 3 months
  Measure respiratory rate using Lifelight® with tolerance accuracy closer to 100% of readings within 5 breaths per minute.
Secondary Objective 4 | 3 months
  Measure systolic and diastolic blood pressure using Lifelight® with accuracy closer to 5+/- 8mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Wiffen, Principal Investigator — Portsmouth Hospitals University NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No